CLINICAL TRIAL: NCT02494505
Title: Does the Mycophenolate Improve the Ability of Weaning Patients Off the Treatment in Chronic Inflammatory Demyelinating Polyradiculopathy (CIDP)
Brief Title: Interest of Mycophenolate for CIDP Weaning
Acronym: MYCOPID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P110148
Record Dates: First submitted 2015-06-10; First posted 2015-07-10 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculopathy
Keywords: chronic inflammatory demyelinating polyradiculopathy; intravenous immunoglobulin (IVIG); withdrawal; quality of life; Clinical trial; cost
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mycophenolate mofetil (Experimental)
  Interventions: Drug: Mycophenolate Mofetil
- placebo (Placebo Comparator): placebo pills
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mycophenolate Mofetil — 2g/day per os
  Arms: mycophenolate mofetil
Drug: placebo
  Arms: placebo

SUMMARY:
The main objective is to study if the mycophenolate could decrease the proportion of patients who relapse during the IVIG tapering period and after the IVIG withdrawal.

DETAILED DESCRIPTION:
The secondary objectives are :

* Study if the mycophenolate could improve the proportion of withdrew patients.
* Study if the mycophenolate could improve the reduction of IVIG dose or could prolong the interval between two courses of IVIG compared to the baseline interval at month 12 and month 24 (= sparing treatment criteria).
* Study if mycophenolate could short the delay to perform the IVIG withdrawal.
* Study if mycophenolate could improve the clinical scores (ONLS, R-ODS MRC, INCAT sensory, 10 meters test) or pain score at month 12 and month 24.
* Study if mycophenolate could improve the quality of life at month12 and month 24.
* Identify clinical, biological and electrophysiological factors associated with withdrawal.
* To assess the pharmacokinetics factors (Area under the curve measuring the exposure to mycophenolate) and the pharmacogenetic factors (cytochrome and carrier, FcgammaR) associated with withdrawal.
* Evaluate the tolerance of Mycophenolate in this new indication.

ELIGIBILITY:
Inclusion criteria :

* Patient older than eighteen
* Written informed consent for study participation
* Definite or probable CIDP according to EFNS/PNS criteria or atypical CIDP (need to meet clinical EFNS/PNS criteria and at least 2 criteria among the EFNS/PNS supplementary criteria)
* Being responder (= decrease of at least 1 point on the ONLS score after IVIG) and dependent to IVIG (= increase of at least 1 point on the ONLS score after IVIG withdrawal or during the tapering period)
* Having received at least 3 courses of IVIG
* Negative pregnancy test for women of child-bearing age

Exclusion criteria :

* No social security benefit
* Pregnancy or intention to become pregnant
* Nursing mother
* Recent or active VIH or hepatitis B or C , or lyme infections
* Monoclonal IgM gammapathy with anti MAG antibodies or CANOMAD syndrome
* Neutropenia < 1G/L
* Malignancy during the 10 years before the inclusion
* Patients having received Mycophenolate
* History of allergy to mycophenolate or placebo excipient
* Patients having received immunosuppressive drugs during the 3 months period before the inclusion
* Patients receiving : plasma exchange, magnesium hydroxide, aluminium hydroxide, cholestyramine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
occurrence of a relapse during the tapering off period | up to 18 months
  occurrence of a relapse during the tapering off period (up to 18 months after baseline) or after the withdrawal during the monitoring period.
  (the withdrawal is defined by the ability to reach the last day of IVIG treatment)

SECONDARY OUTCOMES:
Proportion of withdrew patients | 6 months after the withdrawal
Proportion of withdrew patients at the end of the study | 24 months
Sparing treatment (composite criteria) | 24 months
  extension of the mean interval between IVIG courses at month 12 and month 24 compared to baseline, reduction of the total cumulative dose of IVIG at month 12 and month 24 in the mycophenolate group
Time to reach the withdrawal | 24 months
EVA pain score | 12 months
EVA pain score | 24 months
ONLS scale | 12 months
ONLS scale | 24 months
R-ODS scale | 12 months
R-ODS scale | 24 months
MRC scale | 12 months
MRC scale | 24 months
INCAT sensory test | 12 months
INCAT sensory test | 24 months
10 meters test | 12 months
10 meters test | 24 months
SF-36 | 12 months
  Quality of life scale
SF-36 | 24 months
  Quality of life scale
Nottingham scale | 12 months
  Quality of life scale
Nottingham scale | 24 months
  Quality of life scale
global cost | 24 months
  Comparison of the global cost in each group

CONTACTS AND LOCATIONS:
Overall Officials: Karine Viala, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Neurology - pitié salpetrière hospital, Paris, France